CLINICAL TRIAL: NCT02845128
Title: Prospective Validation of the ROX Index Utility in Predicting Failure of HFNC Treatment in Patients With Acute Respiratory Failure
Brief Title: Prospective Validation of the ROX Index
Status: Completed | Type: Observational
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PR(AG)206/2016
Record Dates: First submitted 2016-07-05; First posted 2016-07-27 (Estimated); Last update posted 2019-08-12 (Actual); Status verified 2018-03

CONDITIONS: Validation
Keywords: high-flow nasal cannula, HFNC, acute respiratory failure, intubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HFNC failure: requiring intubation and invasive mechanical ventilation
- HFNC success: not requiring intubation nor invasive mechanical ventilation

SUMMARY:
We recently described the ROX index, defined as the ratio of SpO2/FIO2 to respiratory rate that outperformed the diagnostic accuracy of the two variables separately. Patients who had a ROX index ≥4.88 after 12 hours of HFNC therapy were less likely to be intubated, even after adjusting for potential covariates. Like any other scoring system, an independent validation of the score in a different population is necessary. We therefore undertook a multicenter, prospective study to validate the ROX index's diagnostic accuracy for determining which patients will fail on HFNC and will need to be intubated.

DETAILED DESCRIPTION:
A growing interest in the non-invasive management of acute respiratory failure has been fuelled by the advent of high-flow nasal canula oxygen therapy (HFNC) and recent data showing that use of HFNC was associated with lower mortality, more ventilator-free days and lower risk for intubation in subsets of patients with PaO2/FIO2≤200mmHg or in those who were immunocompromised in comparison with non-invasive ventilation or standard oxygen. These positive results in favour of HFNC followed physiological studies indicating oxygenation and comfort improvements associated with HFNC use. This has led clinicians to try this technique in the most severe respiratory failure patients, those with ARDS.

Consubstantial to the increasing use of HFNC is the risk of delaying intubation. This is a major concern since a large body of evidence has shown that patients that fail non-invasive ventilatory management of de novo acute respiratory failure (ARF) have a worse outcome.

The variability in both the decision to intubate and its timing reported in several studies suggest that clinical parameters such as respiratory parameters alone are not sufficient and that the progression of the respiratory failure is not sufficiently taken into account. To address this need, we investigated a new score to identify patients at risk of intubation to help clinicians, with three goals simple to use, accurate, and immediately performable at the patients' bedside by any staff.

ELIGIBILITY:
Inclusion Criteria:

- All consecutive patients admitted to the ICU with pneumonia and treated with HFNC were included

Exclusion Criteria:

* Patients younger than 18 years old
* Patients with indication for immediate intubation
* Patients with limitation of therapeutic effort
* Patients electively intubated for diagnostic or therapeutic procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the ICU with pneumonia and treated with HFNC were included
Sampling Method: Non-Probability Sample
Enrollment: 191 (Actual)
Dates: Start 2016-05; Primary Completion 2017-05 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
HFNC failure | Through study completion (an average of 60 days)
  HFNC failure was defined as need for invasive mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Oriol Roca, MD PhD, Study Director — Vall d'Hebron University Hospital
Locations (5):
- France (2):
  - Hôpital Antoine Béclère, Service de Réanimation polyvalente et surveillance continue, Clamart
  - Hôpital Louis Mourier, Service de Réanimation Médico-Chirurgicale, Colombes
- Spain (3):
  - Hospital Universitari Vall d'Hebron. Universitat Autonoma de Barcelona, Barcelona
  - Hospital del Mar, Barcelona
  - Virgen de la Salud University Hospital, Toledo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roca O, Messika J, Caralt B, Garcia-de-Acilu M, Sztrymf B, Ricard JD, Masclans JR. Predicting success of high-flow nasal cannula in pneumonia patients with hypoxemic respiratory failure: The utility of the ROX index. J Crit Care. 2016 Oct;35:200-5. doi: 10.1016/j.jcrc.2016.05.022. Epub 2016 May 31. PMID 27481760
- [Background] Frat JP, Ragot S, Coudroy R, Constantin JM, Girault C, Prat G, Boulain T, Demoule A, Ricard JD, Razazi K, Lascarrou JB, Devaquet J, Mira JP, Argaud L, Chakarian JC, Fartoukh M, Nseir S, Mercat A, Brochard L, Robert R, Thille AW; REVA network. Predictors of Intubation in Patients With Acute Hypoxemic Respiratory Failure Treated With a Noninvasive Oxygenation Strategy. Crit Care Med. 2018 Feb;46(2):208-215. doi: 10.1097/CCM.0000000000002818. PMID 29099420
- [Background] Frat JP, Thille AW, Mercat A, Girault C, Ragot S, Perbet S, Prat G, Boulain T, Morawiec E, Cottereau A, Devaquet J, Nseir S, Razazi K, Mira JP, Argaud L, Chakarian JC, Ricard JD, Wittebole X, Chevalier S, Herbland A, Fartoukh M, Constantin JM, Tonnelier JM, Pierrot M, Mathonnet A, Beduneau G, Deletage-Metreau C, Richard JC, Brochard L, Robert R; FLORALI Study Group; REVA Network. High-flow oxygen through nasal cannula in acute hypoxemic respiratory failure. N Engl J Med. 2015 Jun 4;372(23):2185-96. doi: 10.1056/NEJMoa1503326. Epub 2015 May 17. PMID 25981908
- [Derived] Roca O, Caralt B, Messika J, Samper M, Sztrymf B, Hernandez G, Garcia-de-Acilu M, Frat JP, Masclans JR, Ricard JD. An Index Combining Respiratory Rate and Oxygenation to Predict Outcome of Nasal High-Flow Therapy. Am J Respir Crit Care Med. 2019 Jun 1;199(11):1368-1376. doi: 10.1164/rccm.201803-0589OC. PMID 30576221